CLINICAL TRIAL: NCT02275013
Title: Levosimendan Administration and Outcome in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Sander, Univ-Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: ea1-044-13b
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Treatment of Left Heart Insufficiency in an Operative Setting of Cardiac Surgery
MeSH Terms: interventions — Simendan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Early: Levosimendan administration within first hour of post-operative ICU admission
  Interventions: Drug: Levosimendan
- Late: Levosimendan administration within 24 hours of post-operative ICU admission but after first hour
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan

SUMMARY:
To assess the effects on outcome of levosimendan with respect to timing of its administration on the postoperative course of high-risk cardiac surgery patients in a retrospective observational study.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery between 2006 and 2013
* levosimendan administration within 24 hours of postoperative ICU admission

Exclusion Criteria:

* patients younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2006-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | until discharge, an average of 3 weeks length of stay
1 year follow-up mortality | 1 year after surgery

SECONDARY OUTCOMES:
Duration of mechanical ventilation | until discharge, an average of 3 weeks length of stay
Incidence of renal dysfunction | until discharge, an average of 3 weeks length of stay
Incidence of renal replacement therapy | until discharge, an average of 3 weeks length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Medicine, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Treskatsch S, Balzer F, Geyer T, Spies CD, Kastrup M, Grubitzsch H, Wernecke KD, Erb JM, Braun JP, Sander M. Early levosimendan administration is associated with decreased mortality after cardiac surgery. J Crit Care. 2015 Aug;30(4):859.e1-6. doi: 10.1016/j.jcrc.2015.03.008. Epub 2015 Mar 13. PMID 25837801